CLINICAL TRIAL: NCT02009670
Title: SCFA Production and Their Metabolic Effects After Inulin Ingestion
Brief Title: Inulin,SCFA Production and Metabolic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Inulin and SCFA production
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13C inulin (Experimental): 13C inulin combined with an inulin load are administered orally
  Interventions: Dietary Supplement: 13C inulin
- Placebo (Placebo Comparator): A placebo is administered orally
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 13C inulin — Oral 13C inulin
  Arms: 13C inulin
Other: Placebo — Oral maltodextrin
  Arms: Placebo

SUMMARY:
In this placebo controlled, double-blind, randomized crossover study the investigators will investigate in overweight/obese healthy male volunteers whether inulin administration will increase intestinal SCFA production, thereby investigating whether this will lead to acute metabolic effects.

DETAILED DESCRIPTION:
Gut microbiota is being increasingly recognized as an important factor in fat distribution, insulin sensitivity and glucose and lipid metabolism. Accordingly, the intestinal microbiota could play an important role in the development of obesity and type 2 diabetes mellitus. The role of gut-derived short-chain fatty acids (SCFA), the formation of which is enhanced by microbial fermentation of fibre, is still controversial. At the present time, our understanding of the effects of SCFA on human metabolism (in gut or systemically) is still limited. The investigators hypothesize that the ingested prebiotic inulin is fermented into SCFA and these SCFA have metabolic effects.

ELIGIBILITY:
Inclusion Criteria:

* Overweight, obese men

Exclusion Criteria:

* athletes
* diabetes mellitus

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Fat oxidation, energy expenditure | 1 study day for each administration
  Fat oxidation and energy expenditure are measured after inulin ingestion

SECONDARY OUTCOMES:
Hormones that influence substrate and energy metabolism | 1 study day for each administration
  Insulin, GLP-1, PYY will be measured in plasma after inulin ingestion
Circulating metabolites | 1 study day for each administration
  Glucose, FFA, TG will be measured in plasma after inulin ingestion
Appetite VAS scoring | 1 study day for each administration
  Visual Analogue Scale for hunger and appetite are completed after inulin ingestion
SCFAs | 1 study day for each administration
  SCFA content (acetate, butyrate and propionate, unlabeled and 13C-labeled) are measured after inulin ingestion in plasma, faeces
Breath sampling 13CO2 | 1 study day for each administration
  In breath samples 13CO2 will be measured after inulin ingestion

CONTACTS AND LOCATIONS:
Overall Officials: CHC Dejong, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] van der Beek CM, Canfora EE, Kip AM, Gorissen SHM, Olde Damink SWM, van Eijk HM, Holst JJ, Blaak EE, Dejong CHC, Lenaerts K. The prebiotic inulin improves substrate metabolism and promotes short-chain fatty acid production in overweight to obese men. Metabolism. 2018 Oct;87:25-35. doi: 10.1016/j.metabol.2018.06.009. Epub 2018 Jun 25. PMID 29953876